CLINICAL TRIAL: NCT02788396
Title: The Impact of Post Stenting Balloon Dilatation on Coronary Microcirculation in ST Segment Elevation Myocardial Infarction (STEMI) Patients Undergoing Primary Percutaneous Coronary Intervention (PPCI)
Brief Title: The Impact of Post Stenting Balloon Dilatation on Coronary Microcirculation in STEMI Patients Undergoing PPCI
Acronym: POSTDILSTEMI
Status: Completed | Type: Observational
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Other Study IDs: B853
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: ST-elevation Myocardial Infarction (STEMI)
Keywords: STEMI; PPCI; post-dilatation; coronary microcirculation
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to assess the impact of NC balloon post-dilatation on coronary microcirculation in patients with ST segment elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PPCI).

DETAILED DESCRIPTION:
Suboptimal stent deployment can lead to future stent failure. Thus, optimising stent deployment with non-compliant balloons (NC balloon) post dilatation (PD) at high pressures is an established strategy. In the context of ST segment elevation myocardial infarction (STEMI), PD has been correlated anecdotally with the no reflow phenomenon.

This study aims to determine the impact of stent post-dilation (PD) with NC balloons at high pressures on coronary microcirculation during PPCI by measuring the index of microcirculatory resistance (IMR) pre and post stent post-dilatation. Pre and post PD, an optical coherence tomography (OCT) study will be performed to assess stent deployment and identify parameters that predict the changes in IMR.

ELIGIBILITY:
Inclusion Criteria

* >18 years of age
* Acute symptoms onset with duration > 20 minutes
* ST-segment elevation ≥ 0.1 mV in ≥ 2 contiguous leads, signs of a true posterior infarction or documented newly developed left bundle branch block
* Infarct related artery with a diameter above 2.5 mm
* Operator's intention to proceed to stent deployment (i.e. not refer for CABG or defer PCI)

Exclusion Criteria

* < 18 year of age
* Symptoms duration > 12 hours
* Unable to give informed consent
* Previous bypass graft surgery
* Previous myocardial infarction
* Pregnancy
* Known severe chronic kidney disease (creatinine clearance ≤30 mL/min), unless the patient is on dialysis
* Unable to receive antiplatelets or anticoagulation (i.e. coagulation disorders, bleeding etc.)
* Haemodynamic instability
* Severe LMS disease
* Culprit vessel diameter < 2.5 mm
* Contraindications to adenosine
* Any study lesion characteristic resulting in the expected inability to deliver OCT catheter to the lesion pre and post PD (e.g. moderate or severe vessel calcification or tortuosity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI patients undergoing PPCI
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Delta index of microcirculatory resistance (dIMR) | index procedure
  Delta index of microcirculatory resistance (dIMR) [dΙΜΡ = IMR post post-dilation (post IMR) - IMR pre post-dilation (pre IMR)]

SECONDARY OUTCOMES:
Minimum stent area (MSA) | index procedure
  Pre and post dilatation minimum stent area
Stent expansion | index procedure
  Pre and post dilatation stent expansion; defined as the minimum stent area divided by the average of proximal and distal reference lumen areas x 100
Stent mal-apposition | index procedure
  Stent mal-apposition pre and post dilatation; defined as a distance between the strut's luminal edge and luminal vessel wall of greater >200 μm for a length >600 μm (appreciable in >3 contiguous frames at a pull-back speed of 20 mm/sec
Intra-stent plaque protrusion and thrombus | index procedure
  Pre and post dilatation intra-stent plaque protrusion and thrombus; defined as a mass attached to the luminal surface or floating within the lumen at least 200 μm beyond the luminal edge of a strut
Stent edge dissections | index procedure
  Edge dissections pre and post dilatation, further defined as major and minor [major dissections defined as the ones with a dissection flap width greater or equal to 200 μm)

CONTACTS AND LOCATIONS:
Overall Officials: John R Davies, MD PhD, Study Chair — Mid and South Essex NHS Foundation Trust
Locations (1):
- The Essex Cardiothoracic Centre, Basildon, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karamasis GV, Kalogeropoulos AS, Gamma RA, Clesham GJ, Marco V, Tang KH, Jagathesan R, Sayer JW, Robinson NM, Kabir A, Aggarwal RK, Kelly PA, Prati F, Keeble TR, Davies JR. Effects of stent postdilatation during primary PCI for STEMI: Insights from coronary physiology and optical coherence tomography. Catheter Cardiovasc Interv. 2021 Jun 1;97(7):1309-1317. doi: 10.1002/ccd.28932. Epub 2020 Apr 23. PMID 32329200